CLINICAL TRIAL: NCT00913198
Title: A Phase II Study of CP-4126 in Patients With Advanced Pancreatic Cancer.
Brief Title: A Study of CP-4126 in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4126-201
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Advanced Adenocarcinoma of Pancreas
Keywords: Pancreas; Advanced adenocarcinoma; CP-4126
MeSH Terms: interventions — CP 4126

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV CP-4126 (Experimental)
  Interventions: Drug: IV CP-4126

INTERVENTIONS:
Drug: IV CP-4126 — 1250 mg/m2/d, IV (in the vein) on day 1, 8 and 15 of each 4 week cycle. Number of Cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The main objective of this study is to assess the biological activity of CP-4126 in patients with advanced pancreatic cancer. In addition, the correlation between hENT1 (human equilibrative nucleoside transporter 1) and overall survival will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed advanced pancreatic cancer*
* Not eligible for curative resection
* Performance Status (ECOG) 0-2
* Estimated life expectancy of at least 12 weeks
* Age ≥ 18 years
* Adequate haematological and biological functions:

  * Neutrophils ≥ 1.5 x 109/L
  * Platelets > 100.0 x 109/L
  * Hb ≥ 10 g/dL
  * AST/ALT and alkaline phosphatase (ALP) ≤ 2.5 x institutional upper limit of normal (ULN), if liver metastases
  * AST/ALT ≤ 5 x institutional ULN and ALP ≤ 4 x institutional ULN
  * Bilirubin ≤ 1.5 times institutional ULN, if liver metastases ≤ 3 x institutional ULN
  * Serum creatinine ≤ 1.5 times institutional ULN
* Signed informed consent

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Symptomatic brain metastases
* Participation in another therapeutic clinical study within 30 days of enrolment or during this clinical study
* Requirement of concomitant treatment with a non-permitted medication, including high doses of vitamins and alternative drugs
* History of allergic reactions to gemcitabine or egg
* Presence of any serious concomitant systemic disorders incompatible with the clinical study (e.g. uncontrolled inter-current illness including ongoing or active infection)
* Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance
* Pregnant or breastfeeding women
* Absence of adequate contraception for both male and female fertile patients for the duration of the study; and also for three months after last treatment
* Known positive status for HIV
* Any reason why, in the investigator's opinion, the patient should not participate in the study.
* Drug or alcohol abuse
* Prior radical resection, but exploratory laparotomy as well palliative (e.g bypass) surgery are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Biological activity of CP-4126 in patients with advanced pancreatic cancer. | Every second cycle

SECONDARY OUTCOMES:
Overall survival, Objective response rate. | Every second cycle - study length

CONTACTS AND LOCATIONS:
Locations (3):
- Clinique d'Oncologie Médicale, Institut Jules Bordet, Brussels, Belgium
- Norway (2):
  - Oslo University Hospital, The Norwegian Radium Hospital,, Oslo
  - Oslo University Hospital, Ullevål, Oslo